CLINICAL TRIAL: NCT00182468
Title: If, When and How to Ask the Question(s): Assessing Screening Approaches to Identifying Woman Abuse in Health Care Settings
Brief Title: Does Routine Screening for Intimate Partner Violence Against Women in Health Care Settings do More Good Than Harm?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Echo: Improving Women's Health in Ontario (formerly Ontario Women's Health Council) (Unknown)
Responsible Party: Dr. Harriet L. MacMillan, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: MacMillan_VAW_RCT
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2009-09-09 (Estimated); Status verified 2009-09

CONDITIONS: Intimate Partner Violence Against Women
Keywords: Domestic violence; Spouse Abuse
MeSH Terms: interventions — Mass Screening

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Women are screened for intimate partner violence prior to seeing a health care provider.
  Interventions: Other: Screening for intimate partner violence
- 2 (No Intervention): Women see their health care provider without being asked about intimate partner violence.

INTERVENTIONS:
Other: Screening for intimate partner violence — Women are screened for intimate partner violence prior to seeing a health care provider.
  Arms: 1

SUMMARY:
The purpose of the research is to evaluate whether routine screening for woman abuse in health care settings, as compared to no screening, does more good than harm. Recent reviews have identified the need for high quality research to understand 1) the actual impact on all women of instituting mass screening procedures to identify woman abuse and 2) the extent to which early identification through screening is effective in preventing or ameliorating important outcomes. The main outcomes for the study are reduction in violence, improvement in life quality, and potential harms of screening. A number of secondary outcomes to help understand the process by which screening and usual care might lead to changes in the primary outcomes will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-64 years
* Patients at the health care site
* Able to participate in English
* Able to separate from accompanying person(s)

Exclusion Criteria:

* Too ill to participate
* Unable to separate from accompanying person(s)
* Unable to speak, read, or write English

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5681 (Actual)
Dates: Start 2005-04; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Recurrence of intimate partner violence | 18 months
Health-specific quality of life | 18 months
Harms of screening and/or usual care | 18 months

SECONDARY OUTCOMES:
Mental health (depression, post-traumatic stress disorder [PTSD], anxiety, somatic complaints, substance use) | 18 months
Global physical and emotional health and well-being | 18 months
Health services utilization | 18 months
Safety behaviours | 18 months
Use of information and resources | 18 months
Child quality of life | 18 months
Stage in process of identifying and resolving abuse | 18 months
Exposure to maltreatment as a child | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Harriet L MacMillan, MD, MSc, Principal Investigator — McMaster University
Locations (28):
- Canada (28):
  - Brantford Aboriginal Health Centre, Brantford, Ontario
  - Joseph Brant Hospital, Burlington, Ontario
  - Sudbury Family Physicians, Greater Sudbury, Ontario
  - Sudbury Brady Clinic, Greater Sudbury, Ontario
  - Sudbury District Health Unit, Greater Sudbury, Ontario
  - Hopital Regional de Sudbury Regional Hospital, Emergency Services, Greater Sudbury, Ontario
  - Grimsby Medical Associates, Grimsby, Ontario
  - West Lincoln Memorial Hospital, Grimsby, Ontario
  - St. Joseph's Centre for Ambulatory Health Services, Hamilton, Ontario
  - Rosedale Medical Group, Hamilton, Ontario
  - North Hamilton Community Health Centre, Hamilton, Ontario
  - Aboriginal Health Centre, Hamilton, Ontario
  - McMaster University Medical Centre, Hamilton, Ontario
  - Hamilton Urban Core Community Health Centre, Hamilton, Ontario
  - City of Hamilton Public Health and Community Services Department, Hamilton, Ontario
  - West End Clinic, Hamilton, Ontario
  - HART Clinic, Hamilton, Ontario
  - Victoria Hospital, London, Ontario
  - St. Joseph's Health Care - Women's Ambulatory Health Centre, London, Ontario
  - St. Joseph's Urgent Care, London, Ontario
  - University Hospital, London, Ontario
  - London Family Practice - Dr. Bhayana, London, Ontario
  - St. Joseph's Family Medical & Dental Centre, London, Ontario
  - Willett Hospital Urgent Care, Paris, Ontario
  - Niagara Health Prompt Care, St. Catharines, Ontario
  - Mt. Sinai Hospital, Obstetrics & Gynecology Clinic, Toronto, Ontario
  - Mt. Sinai Hospital, Toronto, Ontario
  - Central Toronto Community Health Centre, Toronto, Ontario

REFERENCES:
- [Derived] MacMillan HL, Wathen CN, Jamieson E, Boyle MH, Shannon HS, Ford-Gilboe M, Worster A, Lent B, Coben JH, Campbell JC, McNutt LA; McMaster Violence Against Women Research Group. Screening for intimate partner violence in health care settings: a randomized trial. JAMA. 2009 Aug 5;302(5):493-501. doi: 10.1001/jama.2009.1089. PMID 19654384